CLINICAL TRIAL: NCT07344025
Title: Comparative Analysis of Healing Outcomes Between Two Bone Graft Materials in Socket Preservation Procedure
Brief Title: Comparative Analysis of 2 Bone Graft Materials in Socket Preservation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pharos University in Alexandria (Other)
Responsible Party: Principal Investigator, Haitham Sakr, Principle investigator, Pharos University in Alexandria
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PharosU
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Socket Preservation; Alveolar Ridge Augmentation; Dental Implants
Keywords: Alveolar ridge preservation; Allograft; Bovine xenograft

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allograft Group (Experimental): Extraction sockets grafted with cortico-cancellous particulate allograft and covered with a collagen membrane.
  Interventions: Procedure: Socket Preservation with Graft Material Allograft
- Xenograft Group (Experimental): Extraction sockets grafted with xenograft material and covered with a collagen membrane.
  Interventions: Procedure: Socket Preservation with Graft Material Allograft

INTERVENTIONS:
Procedure: Socket Preservation with Graft Material Allograft — Socket preservation will be performed after tooth extraction using graft material Allograft or Xenograft according to standard surgical protocol.
  Other Names: Socket Preservation with Graft Material Xenograft

SUMMARY:
Socket preservation procedures after tooth extraction have been designed and implemented to maintain the volume of the bone and gingival tissues, which can decrease following the extraction of the teeth. In this clinical trial we will compare clinically and histologically the effectiveness of two distinct bovine bone graft materials; an allograft and a xenograft, in alveolar ridge preservation procedures following tooth extraction .

DETAILED DESCRIPTION:
Patients who seek socket preservation procedures will be identified and recruited from the out clinic of College of Dentistry. Inclusion criteria will be: systemically healthy, non-smoking patients aged 21-50 years, with no bone metabolism affecting medications, good oral hygiene (full-mouth plaque score <20%), and willingness to participate. Exclusion criteria included stage III/IV periodontitis, active periodontal lesions, acute infection, severely resorbed sockets (buccal bone height <5 mm), smoking >10 cigarettes/day, and pregnancy.

Indications for extraction include caries, failed endodontic treatment, unrestorable teeth, and tooth fracture. All patients underwent full periodontal examination and initial therapy (oral hygiene instructions, scaling, and root planing) at least 4 weeks before surgery. Preoperative CBCT scans will be analyzed for baseline conditions. Reference stents will be fabricated and used to standardize bone dimensional measurements.

Sample size estimation was based on detecting a mean dimensional change in ridge width following 2-3 months of healing. With SD = 10%, α = 0.05, and power = 80%, a minimum of 9 sockets per group (18 total) was deemed adequate.

Surgical Protocol All surgical procedures will be performed under local anesthesia (2% lidocaine with 1:100,000 epinephrine). A sulcular incision will be made with a 15c blade, and atraumatic extraction will be achieved using periotomes, tooth separation, and forceps while preserving the buccal plate. Following thorough socket debridement, the buccolingual ridge width will be measured using a periodontal probe and customized stent.

Patients will be randomly allocated into one of two treatment groups:

Group 1: Allograft group (n=9) Group 2: Xenograft group (n=9) In all cases, graft material will be condensed gently from the apical region. Sockets will be covered with a collagen membrane and closed with 4-0 PTFE sutures.

All patients will receive standard postoperative care including: amoxicillin 500 mg TID for 7 days, ibuprofen 600 mg BID, and 0.12% chlorhexidine rinse BID for 7 days (starting 48h post-op). Sutures will be removed after 14 days. Patients will be recalled at 2-3 months for CBCT scans with an identical machine and settings. Buccolingual ridge width and buccal bone thickness will be assessed by superimposing baseline and follow-up scans.

At 3 months, crestal/intrasulcular incisions will be made and flaps elevated for re-entry. Biopsies will be obtained using a 2.0-mm trephine bur (8 mm length) from all grafted sites. A total of 27 biopsies (9 per group) will be collected, coded, and fixed in 10% neutral buffered formalin. Osteotomies will be completed, and implants will be placed per manufacturer protocol.

ELIGIBILITY:
Inclusion Criteria:

* • Systemically healthy individuals

  * Non-smokers
  * Age between 21 and 50 years
  * Indicated for tooth extraction and socket preservation
  * Good oral hygiene (full-mouth plaque score <20%)
  * Willingness to participate and provide informed consent

Exclusion Criteria:

* • Stage III or IV periodontitis

  * Active periodontal or periapical infection
  * Severely resorbed sockets (buccal bone height <5 mm)
  * Smoking more than 10 cigarettes per day
  * Pregnancy
  * Systemic conditions or medications affecting bone metabolism

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in buccolingual ridge width | Baseline to 2-3 months
  Difference in ridge width measured clinically and radiographically between baseline and 2-3 months post-extraction

SECONDARY OUTCOMES:
Histomorphometric outcomes | 2-3 months
  Percentage of new bone formation, residual graft material, and soft tissue/marrow space

CONTACTS AND LOCATIONS:
Overall Officials: H Sakr, PhD, Principal Investigator — Pharos university
Locations (1):
- College of Dentistry, Pharos University, Alexandria, Egypt